CLINICAL TRIAL: NCT06048211
Title: Impact of the Stool Color Scale in the French Health Book on the Detection of Neonatal Cholestasis
Brief Title: Impact of the Stool Color Scale on the Detection of Neonatal Cholestasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2022PI149
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Neonatal Cholestasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Stool color scale — observationnal trial about the use of the stool color scale by the health professionnals

SUMMARY:
The stool color scale was set in 2018 in the health books of French children. The study aim is to see if the scale is usefull for healthcare professionals and if this scale has advanced the detection of neonatal cholestasis.

DETAILED DESCRIPTION:
The first part of the study consist in send a questionnaire to health professionnal to see their use of the stool color scale in the health book of newborn.

The second part of the study is to see the age of children with cholestasis at the date of the first consult with a specialist.

ELIGIBILITY:
Inclusion Criteria:

* cholestasis

Exclusion Criteria:

-

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patient under 12 month with cholestasis who consult or was hospitalized for this reason.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
use of stool color scale | 4 month
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France